CLINICAL TRIAL: NCT05650151
Title: Peri-operative Vitamin D Therapy for Patients With Hepatocellular Carcinoma Receiving Hepatectomy
Brief Title: Peri-operative Vitamin D Therapy for Hepatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202209057RINA; 2022-11-007A (Other: Taipei veterans general hospital)
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Vitamin D Deficiency; Hepatocellular Carcinoma; Perioperative Complication
Keywords: Vitamin d therapy; Hepatocellular Carcinoma; Perioperative Complication
MeSH Terms: conditions — Vitamin D Deficiency; Carcinoma, Hepatocellular | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Experimental)
  Interventions: Dietary Supplement: Vitamin D
- Control group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — 576 000 IU D 5-7 days prior to the surgery and 144 000 IU daily on post-operative day 1-2
  Arms: Vitamin D group
Dietary Supplement: Placebo — An equal volume of medium chain triglyceride (MCT, as placebo) to vitamin D 5-7 days prior to the surgery and on the post-operative day 1-2.
  Arms: Control group

SUMMARY:
The goal of this double-blind, randomized controlled trial is to test the effect of short-term and high-dose vitamin D therapy in patients undergoing hepatectomy for hepatocellular carcinoma.

DETAILED DESCRIPTION:
Participants will receive short-term high dose of vitamin D during perioperative period.

The main questions the study aims to answer are:

1. If vitamin D therapy benefits perioperative care
2. If short-term high dose of vitamin D supplement is safe

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years
* Patients will undergo hepatectomy for hepatocellular carcinoma.

Exclusion Criteria:

* Patients with hypercalcemia, hyperparathyroidism, sarcoidosis, multiple myeloma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Infection rate | Perioperative period
  Diagnosed by clinical presentation and relevant biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Yi Han, PHD, Principal Investigator — National Taiwan University Hospital